CLINICAL TRIAL: NCT01913600
Title: Resolute Integrity US A Postapproval Study of the Medtronic Resolute™ Integrity Zotarolimus-Eluting Coronary Stent System in the Treatment of De Novo Lesions in Native Coronary Arteries With a Reference Vessel Diameter of 2.25 mm to 4.2 mm
Brief Title: Resolute Integrity US Extended Length Sub-Study(RI US XL)
Acronym: RI-US XL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Vascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IP 126 1D
Record Dates: First submitted 2013-07-30; First posted 2013-08-01 (Estimated); Results first posted 2017-11-17 (Actual); Last update posted 2019-05-08 (Actual); Status verified 2019-04

CONDITIONS: Coronary Artery Disease
Keywords: TARGET LESION REVASCULARIZATION (TLR); TARGET VESSEL REVASCULARIZATION (TVR); Coronary Artery Disease; MYOCARDIAL INFARCTION (MI); PERCUTANEOUS CORONARY INTERVENTION (PCI); STENT THROMBOSIS; TARGET LESION FAILURE (TLF)
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Resolute Integrity (Other): Resolute Integrity Stent
  Interventions: Device: Resolute Integrity Stent

INTERVENTIONS:
Device: Resolute Integrity Stent — Drug eluting stent (DES)

SUMMARY:
Prospective, multi-center, non-randomized, single-arm, open-label study to assess the safety and efficacy of the Resolute Integrity Stent for the treatment of de novo lesions in native coronary arteries with a reference vessel diameter (RVD) of 2.25 mm to 4.2 mm in patients who receive extended length stents (34 mm or 38 mm) referred to as the Extended Length Study.

DETAILED DESCRIPTION:
The purpose of this postapproval study is to conduct a prospective, multi-center evaluation of the procedural and clinical outcomes of subjects that are treated with the commercially available 34 mm and 38 mm Medtronic Resolute Integrity Zotarolimus-Eluting Coronary Stent System.

Descriptive statistics and 95% confidence intervals will be calculated for clinically relevant variables as described in a separate statistical analysis plan.

ELIGIBILITY:
General and Angiographic Inclusion Criteria highlights:

* Acceptable candidate for percutaneous coronary intervention (PCI),stenting, and emergency coronary artery bypass graft surgery
* Clinical evidence of ischemic heart disease, stable or unstable angina, silent ischemia and/or positive functional study
* Informed consent
* Patient agrees to comply with specified follow-up evaluations
* Single target lesion or two target lesions located in separate coronary arteries
* De novo lesion(s) in native coronary artery(ies)
* Target lesion(s) ≤ 35 mm in length
* Target vessel(s) have reference vessel diameter 2.25 mm to 4.2 mm

General and Angiographic Exclusion Criteria highlights:

* Within 7 days of index procedure platelet count <100,000 cells/mm³ or >700,000 cells/mm³; White blood cell (WBC) count <3,000 cells/mm³; serum creatinine level >2.5 mg/dl
* Acute Myocardial Infarction (MI) within 72 hrs of the intended trial procedure (QWMI or any elevation of Creatine Kinase-MB (CK-MB) > lab upper limit of normal)
* Previous PCI of target vessel(s) within 9 months prior to the procedure
* Planned PCI of any vessel within 30 days post-index procedure and/or planned PCI of target vessel(s) within 12 months post-index procedure
* History of stroke or Transient Ischemic Attack (TIA) within prior 6 months
* Participating in investigational drug/device study that has not completed primary endpoint or interferes with study endpoints
* Inability to comply with required trial antiplatelet regimen
* Previous stent in target vessel unless it has been at least 9 months since stent placed and target lesion(s) is/are at least 15 mm from previous stent
* Target vessel(s) has/have other lesions w/ > 40% diameter stenosis
* Unprotected left main coronary artery disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- St. Joseph's Hospital Health Center, Syracuse, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 56 XL subjects were enrolled from 9 study sites in the United States. The first subject was enrolled on July 26, 2013 and the last subject was enrolled on October 27, 2015.
Groups:
- Resolute Integrity US Extended Length Sub-Study (RI-US XL): Resolute Integrity Stent
  Resolute Integrity Stent: Drug eluting stent (DES)
  Description - Patients with at least one lesion amendable to treatment with a 34 or 38 mm length stent. For those subjects with a second lesion, the second lesion may be treated with any available size study stent. Subjects treated with a 34mm or 38mm length stent were designated as a participant in the XL sub study regardless of the length of any other stent that was implanted as part of the study procedure.
Period: Overall Study
Arm/Group | Resolute Integrity US Extended Length Sub-Study (RI-US XL)
Started | 56
Completed | 55
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Resolute Integrity US Extended Length Sub-Study (RI-US XL)
Number analyzed (Participants) | 56
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.5 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 43
Region of Enrollment [Number; unit: participants]
  United States | 56

OUTCOME MEASURES:

1. Primary Outcome: Composite Rate of Cardiac Death and Target Vessel Myocardial Infarction (MI)
Description: The combined clinical outcome of (all cause) mortality, MI or any revascularization
Time Frame: 12 months
Population: 2 subjects did not complete the 12 month follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Resolute Integrity US Extended Length Sub-Study (RI-US XL)
Number analyzed (Participants) | 54
Participants | 4

2. Secondary Outcome: Composite Endpoint: Major Adverse Cardiac Events (MACE)
Description: Defined as death, myocardial infarction (Q wave and non-Q wave), emergent coronary bypass surgery, or clinically-driven repeat target lesion revascularization by percutaneous or surgical methods.
Time Frame: 30 days, 6 months, 12 months
Population: 2 subjects did not complete the 12 month follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Resolute Integrity US Extended Length Sub-Study (RI-US XL)
Number analyzed (Participants) | 56
Participants
  30 Days | 2
  180 Days | 2
  360 Days: number analyzed (Participants) | 54
  360 Days | 5

3. Secondary Outcome: Composite Endpoint: Target Lesion Failure (TLF)
Description: Defined as cardiac death, target vessel myocardial infarction (Q wave and non-Q wave), or clinically-driven target lesion revascularization (TLR) by percutaneous or surgical methods
Time Frame: 30 days, 6 months, 12 months
Population: 2 subjects did not complete the 12 month follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Resolute Integrity US Extended Length Sub-Study (RI-US XL)
Number analyzed (Participants) | 56
Participants
  30 Days | 2
  180 Days | 2
  360 Days: number analyzed (Participants) | 54
  360 Days | 4

4. Secondary Outcome: Composite Endpoint: Target Vessel Failure (TVF),
Description: The composite endpoint comprised of cardiac death, target vessel myocardial infarction, or clinically-driven target vessel revascularization by percutaneous or surgical methods.
Time Frame: 30 days, 6 months, 12 months
Population: 2 subjects did not complete the 12 month follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Resolute Integrity US Extended Length Sub-Study (RI-US XL)
Number analyzed (Participants) | 56
Participants
  30 Days | 2
  180 Days | 2
  360 Days: number analyzed (Participants) | 54
  360 Days | 4

5. Secondary Outcome: Composite Endpoint: Cardiac Death and Target Vessel MI
Description: Combined rate of cardiac death and target vessel MI post-procedure
Time Frame: 30 days, 6 months, 12 months
Population: 2 subjects did not complete the 12 month follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Resolute Integrity US Extended Length Sub-Study (RI-US XL)
Number analyzed (Participants) | 56
Participants
  30 Days | 2
  180 Days | 2
  360 Days: number analyzed (Participants) | 54
  360 Days | 4

6. Secondary Outcome: Composite Endpoint: Target Vessel MI
Description: Target-vessel MI is defined as a MI that occurs in a territory that cannot be clearly attributed to a vessel other than the target vessel.
Time Frame: 30 days, 6 months, 12 months
Population: 2 subjects did not complete the 12 month follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Resolute Integrity US Extended Length Sub-Study (RI-US XL)
Number analyzed (Participants) | 56
Participants
  30 Days | 2
  180 Days | 2
  360 Days: number analyzed (Participants) | 54
  360 Days | 3

7. Secondary Outcome: Clinical Endpoint: Death
Description: All deaths including cardiac death, vasular death and non-cardiovascular death
Time Frame: 30 days, 6 months, 12 months
Population: 2 subjects did not complete the 12 month follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Resolute Integrity US Extended Length Sub-Study (RI-US XL)
Number analyzed (Participants) | 56
Participants
  30 Days | 0
  180 Days | 0
  360 Days: number analyzed (Participants) | 54
  360 Days | 1

8. Secondary Outcome: Clinical Endpoint: Myocardial Infarction (MI)
Description: All myocardial infarction data will be reported per Medtronic historical protocol definitions and according the Academic Research Consortium (ARC) definitions.
Time Frame: 30 days, 6 months, 12 months
Population: 2 subjects did not complete the 12 month follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Resolute Integrity US Extended Length Sub-Study (RI-US XL)
Number analyzed (Participants) | 56
Participants
  30 Days | 2
  180 Days | 2
  360 Days: number analyzed (Participants) | 54
  360 Days | 4

9. Secondary Outcome: Clinical Endpoint: Target Lesion Revascularization (TLR)
Description: Repeat Percutaneous coronary intervention (PCI) or Coronary artery bypass grafting (CABG) to the target lesion.
Time Frame: 30 days, 6 months, 12 months
Population: 2 subjects did not complete the 12 month follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Resolute Integrity US Extended Length Sub-Study (RI-US XL)
Number analyzed (Participants) | 56
Participants
  30 Days | 0
  180 Days | 0
  360 Days: number analyzed (Participants) | 54
  360 Days | 1

10. Secondary Outcome: Clinical Endpoint: Target Vessel Revascularization (TVR)
Description: Repeat PCI or CABG of the target vessel.
Time Frame: 30 days, 6 months, 12 months
Population: 2 subjects did not complete the 12 month follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Resolute Integrity US Extended Length Sub-Study (RI-US XL)
Number analyzed (Participants) | 56
Participants
  30 Days | 0
  180 Days | 0
  360 Days: number analyzed (Participants) | 54
  360 Days | 1

11. Secondary Outcome: Clinical Endpoint: Stent Thrombosis
Description: All stent thrombosis data will be reported per Medtronic historical protocol definitions and according the Academic Research Consortium (ARC) definitions
Time Frame: Early Thrombosis (<=30 days), Late Thrombosis (31-360 days)
Population: 2 subjects did not complete the 12 month follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Resolute Integrity US Extended Length Sub-Study (RI-US XL)
Number analyzed (Participants) | 56
Participants
  Early Thrombosis (<=30 days): number analyzed (Participants) | 54
  Early Thrombosis (<=30 days) | 1
  Late Thrombosis (31-360 days): number analyzed (Participants) | 54
  Late Thrombosis (31-360 days) | 0

12. Secondary Outcome: Clinical Endpoint: Stroke
Description: Defined as sudden onset of vertigo, numbness, dysphasia, weakness, visual field defects, dysarthria or other focal neurological deficits due to vascular lesions of the brain such as hemorrhage, embolism, thrombosis, or rupturing aneurysm, that persists more than 24 hours.
Time Frame: 30 days, 6 months, 12 months
Population: 2 subjects did not complete the 12 month follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Resolute Integrity US Extended Length Sub-Study (RI-US XL)
Number analyzed (Participants) | 56
Participants
  30 Days | 0
  180 Days | 0
  360 Days: number analyzed (Participants) | 54
  360 Days | 0

13. Secondary Outcome: Clinical Endpoint: Bleeding Complications in General
Description: Bleeding complications in general including the GUSTO classification of Severe, Moderate & Mild will be collected. The GUSTO scale defines clinical events that stratify bleeding episodes into mild, moderate or severe.
Time Frame: 30 days, 6 months, 12 months
Population: 2 subjects did not complete the 12 month follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Resolute Integrity US Extended Length Sub-Study (RI-US XL)
Number analyzed (Participants) | 56
Participants
  30 Days | 3
  180 Days | 6
  360 Days: number analyzed (Participants) | 54
  360 Days | 9

14. Secondary Outcome: Dual Antiplatelet Therapy (DAPT) Compliance
Description: Protocol defined DAPT, Aspirin and Clopidogrel or Ticlopidine, at 30 days, 180 day and 360 days.
Time Frame: 30 days, 6 months, 12 months
Population: At the time of the 12 month follow up there were 52 subjects with evaluable data
Measure: Count of Participants; unit: Participants
Arm/Group | Resolute Integrity US Extended Length Sub-Study (RI-US XL)
Number analyzed (Participants) | 56
Participants
  30 Days | 47
  180 Days | 47
  360 Days: number analyzed (Participants) | 52
  360 Days | 40

ADVERSE EVENTS:
Time Frame: 1 Year
Arm/Group | Resolute Integrity US Extended Length Sub-Study (RI-US XL)
All-Cause Mortality (participants affected / at risk) | 1/56
Serious Adverse Events (participants affected / at risk) | 45/56
Other Adverse Events (participants affected / at risk) | 45/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Resolute Integrity US Extended Length Sub-Study (RI-US XL) (N=56)
Acute MI (Cardiac disorders) | 3
Anaemia (Blood and lymphatic system disorders) | 1
Angina Unstable (Cardiac disorders) | 4
Atrial Fibrilation (Cardiac disorders) | 1
Atrial Flutter (Cardiac disorders) | 1
Cardiac Failure (Cardiac disorders) | 1
Cardiac Failure Congestive (Cardiac disorders) | 2
Coronary Artery Disease (Cardiac disorders) | 2
Coronary Artery Dissection (Cardiac disorders) | 3
Retinal Detachment (Eye disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1
Pancreatitis Acute (Gastrointestinal disorders) | 1
Polyp Colerectal (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 1
Ischaemic Hepatitis (Hepatobiliary disorders) | 1
Bronchitis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Postoperative Wound Infection (Infections and infestations) | 1
Upper Respiratory Tract Infection (Infections and infestations) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Lung Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal Failure Acute (Renal and urinary disorders) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Mass (Respiratory, thoracic and mediastinal disorders) | 1
Hypertension (Vascular disorders) | 2
Hypotension (Vascular disorders) | 1
Intermittent Claudication (Vascular disorders) | 1
Orthostatic Hypotension (Vascular disorders) | 1
Peripheral Arterial Occlusive Disease (Vascular disorders) | 1
Vasospasm (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Resolute Integrity US Extended Length Sub-Study (RI-US XL) (N=56)
Palpitations (Cardiac disorders) | 5
Dyspepsia (Gastrointestinal disorders) | 4
Chest Pain (General disorders) | 11
Fatigue (General disorders) | 4
Bronchitis (Infections and infestations) | 5
Cardiac Enzymes Increased (Investigations) | 8
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No